CLINICAL TRIAL: NCT01162174
Title: Effects of Oligonol on Vascular Function and Inflammation in Healthy Men: A Double-Blind, Dose-Finding Study
Brief Title: Pilot Study of Oligonol Supplementation to Promote Cardiovascular Health
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Amino Up Chemical Company (Industry)
Responsible Party: Carl L Keen, University of California, Davis
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 200816212-1
Record Dates: First submitted 2010-07-12; First posted 2010-07-14 (Estimated); Last update posted 2010-07-14 (Estimated); Status verified 2010-07

CONDITIONS: Cardiovascular Health
Keywords: Flavanols; cardiovascular
MeSH Terms: interventions — oligonol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 100 mg of Oligonol (Experimental)
  Interventions: Dietary Supplement: Oligonol
- 200 mg of Oligonol (Experimental)
  Interventions: Dietary Supplement: Oligonol
- 0 mg of Oligonol (Placebo Comparator)
  Interventions: Dietary Supplement: Oligonol

INTERVENTIONS:
Dietary Supplement: Oligonol

SUMMARY:
The investigators hypothesize that acute consumption of Oligonol, a patented lychee fruit extract (Amino Up Chemical Co.) particularly rich in low molecular weight flavanols, will improve endothelial function, reduce platelet reactivity and increase circulating levels of flavonoids after a single intake.

DETAILED DESCRIPTION:
The investigators have demonstrated from previous studies at UC Davis that a single dose of a high-flavanol supplement from cocoa can improve endothelial function, measured by increased blood flow from peripheral arterial tonometry (PAT), reduce platelet reactivity, and increase circulating levels of flavonoids in the blood. The investigators seek with this proposal to determine if a similar response can be noted with a different high-flavanol supplement in normal, healthy people.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50 yrs.
* Healthy, not taking prescription medications
* Subject is willing and able to comply with the study protocols.
* Subject is willing to consume the Oligonol extract drink or placebo once a week for each of three weeks.

Exclusion Criteria:

* Physical signs of health impairment.
* Abnormal clinical laboratory (CBC, chemistry, liver, etc.) values if determined to be clinically significant by Dr. Eric Gershwin
* Inflammatory disorders (e.g. rheumatoid arthritis)
* Malabsorption
* Treatment with corticosteroids, hypolipidemic and anti-inflammatory drugs
* Renal or Liver disease
* Heart Disease, which includes cardiovascular events and stroke
* Cushing's syndrome
* History of psychiatric disorders i.e. schizophrenia or bi-polar or depression treated with antidepressants within the last 1 year.
* Anti-anxiety medications
* Routine use of prescription drugs or over-the counter medications, which may potentially modulate the outcome of this study; including antibiotics, aspirin and aspirin-containing formulations, COX-2 inhibitors, antihistamines, corticosteroids, ACE-inhibitors, and beta-blockers, erectile dysfunction drugs.
* Asthma (can be worsened by mild to moderate food allergies).
* Indications of substance or alcohol abuse within the last 3 years
* Undergoing nicotine cessation therapy
* Multi-Vitamin and mineral use other than a One-A-Day type formula
* Current, consistent use of herbal or plant-based supplements; omega-3 fatty acids, and fish or unwilling to discontinue use while participating in the study.
* Alcohol consumption > 1 oz/day (2 beers/day or 2 glasses of wine/ day, 1 drink of hard liquor/day)
* Chronic high-intensity exercise
* Smoking

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2008-08; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Peripheral Arterial Tonometry | 0 and 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Hackman, PhD, Principal Investigator — University of California, Davis